CLINICAL TRIAL: NCT05436080
Title: Epididymal Ultrasongraphic Findings in Asthenozoospermic Infertile Men and Correlation With Seminal Parameters and L.Carnitine Level
Brief Title: Epididymal U.S Findings in Asthenozoospermic &Correlation With L.Carnitine Level
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Abo Elyamen, Dr, Assiut University
Other Study IDs: epididymal findindgs by u.s
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Asthenozoospermia
MeSH Terms: conditions — Asthenozoospermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: U/S — Epididymal Ultrasongraphic Findings by Scrotal U/S

SUMMARY:
To evaluate the epididymal findings by U.S and study its correlation with seminal parameters including L.carnitine level in infertile males

DETAILED DESCRIPTION:
infertility is a relatively common problem affecting about15-20% of reproductive aged couples. Historically, the cause of infertility was falsified attributed to the female partner, while the male factor, which is either primary or a co factor in 40-60% of cases, has largely been ignored Thus, it is important to evaluate men at the same time with women.(2) The epididymis is an elongated structure, posterolateral to the testis within the scrotal sac. Its primary function is the collection, maturation and transport of sperm from rete testis to the ductus deferens.(1)(3) Testicular spermatozoa are nonfunctional and lack the ability to naturally fertilize an oocyte .After, spermatozoa reach the epididymis they undergo a complicated maturation process leading to biochemical, physiological and functional changes resulting in a functional spermatozo on that is able to successfully fertilize an oocyte (3)(4)(8) Sperm dysfunctions are recognised as the most significant cause of male infertility and many may think that sperm dysfunction is only as a result of defective spermatogenesis. However, it can also be the result of an inadequate epididymal maturation process due to improper epididymal function (6)(7)(8) Scrotal sonography is commonly used for evaluation of the infertile male. While abnormalities of the epididymis like( cysts and calcifications ) are frequently observed during sonographic assessment and their presence has uncertain importance (1)(10)(12)(13) Measurement of acetyl carnitine content of human seminal plasma could be used as a marker of epididymal maturation. Carnitine is present in the epididymis at higher concentrations than in other body tissues in the rat

ELIGIBILITY:
Inclusion Criteria:

* 80 married male( 50 asthenzoospermic infertile male and 30 with normal semen male) Age from 18 to 55 years.

Exclusion Criteria:

* Extreme age
* Single
* Recent L carnitine intake
* Undesended testis
* Genetic cause of inferitility
* Patients with clinical Varicocele
* Azoospermic patients

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — evaluate the epididymal findings by U.S and study its correlation with seminal parameters including L.carnitine level in infertile males.
Study Population: Study participants: Patients will be chosen from those attending the outpatient clinic of department of Dermatology, Venereology and Andrology, Assuit University hospitals
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the percentage of epididymal head echotexture in asthenozoospermic infertile male and study its correlation with seminal parameters and L.carnitine level | Baseline
  The sample size calculation was performed using G.power 3.1.9.2 (Universitat Kiel, Germany). The sample size was calculated as total n ≥65 with an allocation ratio of 5:3 in cases and control groups based on the following considerations: 0.05 α error and 80% power of the study to demonstrate that the percentage of epididymal head echotexture heterogeneity is 60% in infertile men (the primary outcome) compared to 25% in healthy fertile men according to a previous study by (Lotti et al., 2021). 15 cases were added to overcome dropout. Therefore, 80 patients will be allocated as 30 cases in fertile group and 50 cases in infertile group.
  Lotti, F., Frizza, F., Balercia, G., Barbonetti, A., Behre, H. M., Calogero, A. E., et al. 2021. The European Academy of Andrology (EAA) ultrasound study on healthy, fertile men: Scrotal ultrasound reference ranges and associations with clinical, seminal, and biochemical characteristics. Andrology, 9, 559-576

SECONDARY OUTCOMES:
Evaluate other epididymal ultrasongraphic findings and study its correlation with seminal parameters and L.carnitine level | Baseline
  Evaluate other epididymal ultrasongraphic findings like( vascularity ,cyst, volume) and study its correlation with seminal parameters and L.carnitine level

CONTACTS AND LOCATIONS:
Overall Officials: Emad abdel rahiem taha, Study Director — Assiut University; Ahmed mahmoud el shibany, Study Director — Assiut University

REFERENCES:
- [Background] Lotti F, Frizza F, Balercia G, Barbonetti A, Behre HM, Calogero AE, Cremers JF, Francavilla F, Isidori AM, Kliesch S, La Vignera S, Lenzi A, Marcou M, Pilatz A, Poolamets O, Punab M, Peraza Godoy MF, Rajmil O, Salvio G, Shaeer O, Weidner W, Maseroli E, Cipriani S, Baldi E, Degl'Innocenti S, Danza G, Caldini AL, Terreni A, Boni L, Krausz C, Maggi M. The European Academy of Andrology (EAA) ultrasound study on healthy, fertile men: Scrotal ultrasound reference ranges and associations with clinical, seminal, and biochemical characteristics. Andrology. 2021 Mar;9(2):559-576. doi: 10.1111/andr.12951. Epub 2021 Jan 19. PMID 33244893